CLINICAL TRIAL: NCT03226210
Title: Comparison of Efficacy and Safety of Prandilin and NovoRapid Evaluated by Continuous Glucose Monitoring System in Newly Diagnosed Type 2 Diabetes
Brief Title: Comparison of Efficacy and Safety of Prandilin and NovoRapid in Newly Diagnosed Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIA-THY-2
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Rapid-acting insulin analogues; Continuous glucose monitoring system (CGMS); Continuous subcutaneous insulin infusion (CSII)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NovoRapid group (group Asp) (Experimental)
  Interventions: Drug: aspart insulin or lipro insulin
- Prandilin group (group Lis) (Experimental)
  Interventions: Drug: aspart insulin or lipro insulin

INTERVENTIONS:
Drug: aspart insulin or lipro insulin — After completing OGTTS, enrolled subjects (new diagnosed T2DM) were randomly assigned into two groups: NovoRapid group (group Asp, Novo Nordisk, Bagsvaerd, Denmark) and Prandilin group (group Lis, Gan & Lee pharmaceuticals, Beijing, China) in CSII, combined with metformin (Bristol-Myers Squibb, USA) therapy. During insulin intensive therapy, every patient general use 1.5g metformin per day. If the patient is unable to tolerate the side effects of metformin, such as diarrhea, nausea, vomiting, allergies, etc., the daily dose of metformin is reduced to 1.0g. If the patients are still unable to tolerate the daily 1.0g of metformin, exit from this study.

SUMMARY:
To compare the effect of the rapid-acting insulin analogues (RAIAs) NovoRapid (aspart) and Prandilin (lispro) on glycemic variations by Continuous glucose monitoring system (CGMS) in continuous subcutaneous insulin infusion (CSII) with metformin intensive therapy in newly diagnosed type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The study was designed as a single blind randomized control trial. A total of 110 newly type 2 diabetic diagnosed patients with hemoglobin A1c (HbA1c%) above 9% were hospitalized, and were randomly divided into two groups: NovoRapid group (group Asp) and Prandilin group (group Lis) in CSII, combined with metformin therapy. Treatments were maintained for 2-3 weeks after the glycaemic target was reached. To complete the assessment of general information, fasting C-peptide (C-P0), 2-h postprandial C-peptide (C-P2h), fasting insulin (Ins0), 2-h postprandial insulin (Ins2h), HbA1c% and fructosamine on the baseline and endpoint. 4 days continuous glucose monitoring (CGM) was performed on after three days stable glucose.

ELIGIBILITY:
Inclusion Criteria:

1. voluntary to attend this study signed the informed consent; 2. between 18 and 75 years of age; 3. according to the who standards, the subjects should be newly diagnosed as type 2 diabetes; 4. BMI between 19 and 35kg/m2; 5.HbA1c>9%; 6. using enough contraception and not pregnancy; 7. The patients do not attend any medical subjectsin in the last 3 months before enrollment; 8. the subjects agreed to maintain the original diet and exercise habits throughout the study period.

Exclusion Criteria:

1. Patients with severe cardiopulmonary disease; 2. Patients with acute complications (diabetic ketoacidosis, diabetic ketosis hypertonic coma, diabetes lactic acidosis, etc.); 3. Patients with intolerance to metformin allergy to metformin 4. Patients with history of mental disease, and not suitable for the use of insulin pump; 5. Researchers think that the patients does not fit for this research (such as alcoholism, drug abuse, etc.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the between-group difference of MAGE | 14 days
  the 24-h mean amplitude of glycemic excursions (MAGE)

CONTACTS AND LOCATIONS:
Overall Officials: Bingli Liu, Doctor, Study Director — Nanjing Medical University
Locations (1):
- Nanjing First Hostital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No